CLINICAL TRIAL: NCT04680806
Title: Gingival Depigmentation With Er,Cr:YSGG and Diode Laser: Randomized Clinical Trial to Evaluate the Repigmentation and Patient Perceptions
Brief Title: Laser-Assisted Gingival Depigmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academy of Laser Dentistry - Gulf Laser Chapter (Other)
Collaborators: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GulfLaserChapter
Record Dates: First submitted 2020-12-15; First posted 2020-12-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Hyperpigmentation; Melanin; Laser-Induced Hyperpigmentation
Keywords: Depigmentation; Gingival Hyperpigmentation; Diode laser; Er,Cr:YSGG laser; Repigmentation
MeSH Terms: conditions — Hyperpigmentation; Vitiligo | interventions — Lasers, Semiconductor

STUDY DESIGN:
Intervention Model Description: Participants were randomly allocated to the two treatment groups: -Group A was treated by an Er,Cr:YSGG laser 2780 nm.
  -Group B: was treated with diode 940 nm Laser.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Allocation of the patients into the two treatment groups was carried out using randomization table with allocation ratio 1:1.
  Participants, investigator, the tree external clinical examiners were blinded about the allocation of the patient in the treatment group.
  Care provider didn't interfere in collecting and analysing the data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Er,Cr:YSGG laser 2780 nm (Experimental): Group A was treated by an Er,Cr:YSGG laser 2780 nm cylindrical tip (tip 600 μm, 45 millijoule /pulse, average power 2.25 W, frequency 50 Hz, pulse duration 60 µs, energy density 43 J/cm2, water 50%, and air 40%). The procedure was performed completely without anesthesia with the laser tip at angulation ~30° and distance of ~1 mm from the gingival tissue. The laser tip was advancing in scanning movement from in the cervical-apical direction in all pigmented areas. The following settings was used to achieve hemostasis in case of the bleeding was present (tip 600 μm, 30 millijoule /pulse, average power 1.5 W, frequency 50 Hz, pulse duration 700 µs, energy density 28.7 J/cm2, water 10%, and air 20%).
  Interventions: Device: Er,Cr:YSGG laser 2780 nm
- Diode laser 940 nm (Experimental): Group B was treated with diode 940 nm Laser. The procedure was performed with a pencil-sized handpiece containing a 400 µm lasing fiber (400 μm initiated tip, average power 0.8 watts, Pulsed mode, Duty cycle 20%, Pulse duration 10 μs, energy density 636.9 J/cm2 per second, no water or air). Infiltration anesthesia was injected for B group . The laser tip was placed in angle ~30° with the gingival surface. Short light paint brush strokes were used in the cervical-apical direction in all pigmented areas.
  Interventions: Device: Diode laser 940 nm

INTERVENTIONS:
Device: Er,Cr:YSGG laser 2780 nm — The depigmentation procedure essentially involves laser ablation of epithelial layer of buccal gingiva containing melanin pigmentation.
  Arms: Er,Cr:YSGG laser 2780 nm
Device: Diode laser 940 nm — The depigmentation procedure essentially involves laser ablation of epithelial layer of buccal gingiva containing melanin pigmentation.
  Arms: Diode laser 940 nm

SUMMARY:
This randomized clinical trial evaluated the recurrence rates of physiological gingival pigments during 24 months follow-up and the patient perceptions after the ablative depigmentation using two laser wavelengths; Diode 940 nm and Er,Cr:YSGG 2780 nm.

DETAILED DESCRIPTION:
This study aim to compare the clinical outcomes, the rate of repigmentation, and the patient perceptions after laser-assisted gingival depigmentation with diode 940 nm and Erbium, chromium-doped yttrium, scandium, gallium and garnet (Er,Cr:YSGG) 2780 nm. Two pigmentation index were used to compare between the treatment outcomes of using Diode laser or Er,Cr:YSGG.

The depigmentation procedure essentially involves ablation of epithelial layer of buccal gingiva containing melanin pigmentation.

Sixty healthy patients (22 males and 38 females, aged 21 to 43 years) who presented with a chief complaint of having dark-brown to black gingival hyperpigmentation between April 2015 and September 2018. Participants were randomly divided into 2 groups (30 patients each). Randomization was carried out using randomization table; by a computer-generated randomization list (SPSS v23.0) with allocation ratio 1:1.

All of the patients were selected according to the study inclusion and exclusion criteria.

Data collection was done by a dental specialist who was blinded about the provided treatment. Data collections included the clinical examination at baseline and follow up appointments. To achieve blinding, three calibrated external experts, blinded to the provided treatment classified the degree of gingival pigments and gingival topography according oral pigmentation index (DOPI) and melanin pigmentation index.

The periodontal surgery was performed by a periodontist specialised in laser dentistry. The periodontist did not interfere with the treatment option.

Descriptive statistics and statistical analysis was done by an external expert using SPSS Statistics software(SPSS v23.0) . Nonparametric tests, Kruskal-Wallis test was used to compare between the two groups according the time intervals.

The patients who did not show in all the study follow up's appointments were dropped from the data analysis.

Patients were asked to evaluate the procedure by using a self-administered questionnaire. The patients were recalled after 1 week, 1 month, 12 months and 24 months.

ELIGIBILITY:
Inclusion Criteria:

• All patient exhibiting physiologic pigmentation of score2 or more according to Oral pigmentation index (DOPI)

Exclusion Criteria:

* Pathologic hyperpigmentation
* Participants with a systemic condition that could affect tissue healing (e. g., autoimmune diseases)
* Pregnancy and lactation
* History of smoking
* Previous mucogingival surgery at the region to be treated
* No contraindication for the laser treatment.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-04-05 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2019-10-20 (Actual)

PRIMARY OUTCOMES:
Oral pigmentation index (DOPI) | Baseline
  * Score 1: No clinical pigmentation (pink-colored gingiva)
  * Score 2: Mild clinical pigmentation (mild light brown color)
  * Score 3: Moderate clinical pigmentation (medium brown or mixed pink and brown color)
  * Score 4: Heavy clinical pigmentation (deep brown or bluish black color)
Oral pigmentation index (DOPI) | 1 month post-operative
  * Score 1: No clinical pigmentation (pink-colored gingiva)
  * Score 2: Mild clinical pigmentation (mild light brown color)
  * Score 3: Moderate clinical pigmentation (medium brown or mixed pink and brown color)
  * Score 4: Heavy clinical pigmentation (deep brown or bluish black color)
Oral pigmentation index (DOPI) | 1 year follow-up
  * Score 1: No clinical pigmentation (pink-colored gingiva)
  * Score 2: Mild clinical pigmentation (mild light brown color)
  * Score 3: Moderate clinical pigmentation (medium brown or mixed pink and brown color)
  * Score 4: Heavy clinical pigmentation (deep brown or bluish black color)
Oral pigmentation index (DOPI) | 2 years follow-up
  * Score 1: No clinical pigmentation (pink-colored gingiva)
  * Score 2: Mild clinical pigmentation (mild light brown color)
  * Score 3: Moderate clinical pigmentation (medium brown or mixed pink and brown color)
  * Score 4: Heavy clinical pigmentation (deep brown or bluish black color)
Melanin pigmentation index: | Baseline
  * Score 0: No pigmentation
  * Score 1: Solitary unit(s) of pigmentation in papillary gingiva without extension between neighboring solitary units
  * Score 2: Formation of continuous ribbon extending from neighboring solitary units
Melanin pigmentation index: | 1 month post-operative
  * Score 0: No pigmentation
  * Score 1: Solitary unit(s) of pigmentation in papillary gingiva without extension between neighboring solitary units
  * Score 2: Formation of continuous ribbon extending from neighboring solitary units
Melanin pigmentation index: | 1 year follow-up
  * Score 0: No pigmentation
  * Score 1: Solitary unit(s) of pigmentation in papillary gingiva without extension between neighboring solitary units
  * Score 2: Formation of continuous ribbon extending from neighboring solitary units
Melanin pigmentation index: | 2 years follow-up
  * Score 0: No pigmentation
  * Score 1: Solitary unit(s) of pigmentation in papillary gingiva without extension between neighboring solitary units
  * Score 2: Formation of continuous ribbon extending from neighboring solitary units
Gingival Appearance | 1 month
  * Score 1:Pink vital appearance for the gingiva
  * Score 2: Pale Non-vital appearance for gingiva

SECONDARY OUTCOMES:
Oral Hygiene Index | Baseline
  The Oral Hygiene Index is composed of the combined Debris Index and Calculus index, each of these index is in turn based on 12 numerical determinations representing the amount of debris or calculus found on the buccal and lingual surfaces of each of three segments of each dental arch.
  Criteria for classifying debris 0 No debris or stain present
  1. Soft debris covering not more than one third of the tooth surface, or presence of extrinsic stains without other debris regardless of surface area covered
  2. Soft debris covering more than one third, but not more than two thirds, of the exposed tooth surface.
  3. Soft debris covering more than two thirds of the exposed tooth surface.
Oral Hygiene Index | 1 month post-operative
  The Oral Hygiene Index is composed of the combined Debris Index and Calculus index, each of these index is in turn based on 12 numerical determinations representing the amount of debris or calculus found on the buccal and lingual surfaces of each of three segments of each dental arch.
  Criteria for classifying debris 0 No debris or stain present
  1. Soft debris covering not more than one third of the tooth surface, or presence of extrinsic stains without other debris regardless of surface area covered
  2. Soft debris covering more than one third, but not more than two thirds, of the exposed tooth surface.
  3. Soft debris covering more than two thirds of the exposed tooth surface.
Gingival Index | Baseline
  The Gingival Index (Löe and Silness, 1963) was created for the assessment of the gingival condition and records qualitative changes in the gingiva. It scores the marginal and interproximal tissues separately on the basis of 0 to 3. The criteria are:
  0= Normal gingiva;
  1= Mild inflammation - slight change in color and slight edema but no bleeding on probing; 2= Moderate inflammation - redness, edema and glazing, bleeding on probing; 3= Severe inflammation - marked redness and edema, ulceration with tendency to spontaneous bleeding.
Gingival Index | 1 month post-operative
  The Gingival Index (Löe and Silness, 1963) was created for the assessment of the gingival condition and records qualitative changes in the gingiva. It scores the marginal and interproximal tissues separately on the basis of 0 to 3. The criteria are:
  0= Normal gingiva;
  1= Mild inflammation - slight change in color and slight edema but no bleeding on probing; 2= Moderate inflammation - redness, edema and glazing, bleeding on probing; 3= Severe inflammation - marked redness and edema, ulceration with tendency to spontaneous bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Omar Hamadah, PhD, Study Director — Damascus University
Locations (1):
- Dr. Tamim Dental Polyclinic, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No
there is no plan to make individual participant data (IPD) available

REFERENCES:
- [Result] Simsek Kaya G, Yapici Yavuz G, Sumbullu MA, Dayi E. A comparison of diode laser and Er:YAG lasers in the treatment of gingival melanin pigmentation. Oral Surg Oral Med Oral Pathol Oral Radiol. 2012 Mar;113(3):293-9. doi: 10.1016/j.tripleo.2011.03.005. Epub 2011 Jun 12. PMID 22676819
- [Result] Nammour S, El Mobadder M, Namour M, Namour A, Rompen E, Maalouf E, Brugnera Junior A, Brugnera AP, Vescovi P, Zeinoun T. A Randomized Comparative Clinical Study to Evaluate the Longevity of Esthetic Results of Gingival Melanin Depigmentation Treatment Using Different Laser Wavelengths (Diode, CO2, and Er:YAG). Photobiomodul Photomed Laser Surg. 2020 Mar;38(3):167-173. doi: 10.1089/photob.2019.4672. Epub 2020 Jan 17. PMID 31951510
- [Result] Hegde R, Padhye A, Sumanth S, Jain AS, Thukral N. Comparison of surgical stripping; erbium-doped:yttrium, aluminum, and garnet laser; and carbon dioxide laser techniques for gingival depigmentation: a clinical and histologic study. J Periodontol. 2013 Jun;84(6):738-48. doi: 10.1902/jop.2012.120094. Epub 2012 Sep 24. PMID 23003920